CLINICAL TRIAL: NCT00827307
Title: The Effects of Adjuvant Zoladex Plus Tamoxifen on Breast Density in Pre- or Peri-menopausal Women With Early-stage Breast Cancer
Brief Title: Zoladex Plus Tamoxifen in Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zhejiang Cancer Hospital (Other)
Responsible Party: Yang Hong-Jian, Zong Xiang-Yun, Zhejiang Cancer Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D8666L00002
Record Dates: First submitted 2009-01-21; First posted 2009-01-22 (Estimated); Last update posted 2011-08-08 (Estimated); Status verified 2011-08

CONDITIONS: Mammography; Estrogen; Lipemia; Endometrium; Ultrasonography
Keywords: breast carcinoma; goserelin; Mammographic density
MeSH Terms: conditions — Hyperlipidemias; Breast Neoplasms | interventions — Tamoxifen; Goserelin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Combination (Experimental): In the combination arm, patients receive ZOLADEX 3.6 mg by subcutaneous injection every 4 weeks along with once-daily oral dose of tamoxifen 20 mg.
  Interventions: Drug: Goserelin
- Conctrol (Active Comparator): In the monotherapy arm, patients receive once-daily oral dose of tamoxifen 20 mg.
  Interventions: Drug: tamoxifen

INTERVENTIONS:
Drug: tamoxifen — In the monotherapy arm, patients receive once-daily oral dose of tamoxifen 20 mg.
  Other Names: TAM
  Arms: Conctrol
Drug: Goserelin — In the combination arm, patients receive ZOLADEX 3.6 mg by subcutaneous injection every 4 weeks along with once-daily oral dose of tamoxifen 20 mg
  Other Names: ZOLADEX
  Arms: Combination

SUMMARY:
The purpose of this study is to compare Zoladex plus tamoxifen with tamoxifen alone as adjuvant hormonal therapy in pre- or perimenopausal women with early-stage breast cancer in terms of breast density, estrogen levels, lipidemia, endometrial thickness and ultrasonographic abnormalities.

DETAILED DESCRIPTION:
After the completion of primary treatment(surgery and/or adjuvant chemotherapy, radiotherapy could be given concurrently with study medication), eligible patients will be randomized to receive Zoladex plus tamoxifen or tamoxifen alone. The duration of study medication along with the follow-up will be 18 months, or until disease recurrence,or discontinuation of study therapy (as a result of an adverse event, a patient's request, or an investigator's decision), further treatment will be at investigator's discretion.

During the study period, contralateral mammograms and transvaginal ultrasound will be undertaken at baseline and after 6, 12 and 18 months of study medications. Mammographic density assessment will be undertaken by a single radiologist. Serum measurements including estrogen levels and lipidemia will be obtained at baseline and after 3, 6, 12 and 18 months of study medications.

ELIGIBILITY:
Inclusion Criteria:

* provision of informed consent
* histologically proven HR+ operable invasive breast cancer
* completion of surgery and chemotherapy(if given).
* women defined as pre- or perimenopausal according to all of the following: aged 50 years or younger, at least one menstrual period during the last months.

Exclusion Criteria:

* clinical evidence of metastatic disease
* pregnancy or breast-feeding
* bilateral oophorectomy;
* radiation of the ovaries
* patients who, for whatever reason(eg, confusion, infirmity,alcoholism),are unlikely to comply with trial requirements
* patients whose chemotherapy was started more than 8 weeks after completion of primary surgery or whose chemotherapy was completed more than 8 weeks before starting the study treatment. Chemotherapy, if given, should have been given post-operatively, ie, patients who received neoadjuvant chemotherapy are ineligible
* patients who have not received chemotherapy and whose primary surgery was completed more than 8 weeks before starting the study treatment
* previous hormonal therapy as adjuvant treatment for breast cancer
* patients unwilling to stop taking any drug known to affect sex hormonal status, or in whom it would be inappropriate to stop
* previous history of invasive malignancy within the last 5 years, other than squamous or basal cell carcinoma of the skin or carcinoma in situ of the cervix, adequately cone biopsied
* treatment with a non-approved or experimental drug during 1 month before entry into the study
* history of hypersensitivity to active or inactive excipients of tamoxifen and Zoladex
* history of bleeding diathesis (ie. Disseminated intravascular coagulation, clotting factor deficiency), or long term anticoagulant therapy (other than antiplatelet therapy and low dose warfarin )
* leukopenia and/or thrombocytopenia
* history of ocular fundus diseases
* history of thromboembolic diseases

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2008-06; Primary Completion 2011-06 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Mammographic percentage density at 18months | 18months after enrolled

SECONDARY OUTCOMES:
estrogen levels, lipidemia, endometrial thickness and ultrasonographic abnormalities | 3,6,12,18 months

CONTACTS AND LOCATIONS:
Overall Officials: Hong-Jian Yang, MD., Principal Investigator — Zhejiang Provicial Cancer Hospital; Xiang-Yun Zong, MD., PhD., Principal Investigator — Zhejiang Cancer Hospital
Locations (1):
- Zhejiang Cancer Hospital, Hangzhou, Zhejiang, China

REFERENCES:
- [Derived] Yang H, Zong X, Yu Y, Shao G, Zhang L, Qian C, Bian Y, Xu X, Sun W, Meng X, Ding X, Chen D, Zou D, Xie S, Zheng Y, Zhang J, He X, Sun C, Yu X, Ni J. Combined effects of goserelin and tamoxifen on estradiol level, breast density, and endometrial thickness in premenopausal and perimenopausal women with early-stage hormone receptor-positive breast cancer: a randomised controlled clinical trial. Br J Cancer. 2013 Aug 6;109(3):582-8. doi: 10.1038/bjc.2013.324. Epub 2013 Jul 16. PMID 23860520